CLINICAL TRIAL: NCT03043703
Title: Accuracy of Detection and Reporting of Sleep-disordered Breathing Metrics Determined by the ResMed AirSense 10 in AirView
Brief Title: AirSense 10 AHI Validation Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study has no principal investigator at the moment.
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ES-RDIVal-01
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Cohort study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AirSense 10 AutoSet for Her (Experimental): Treatment for 1 night with ResMed AirSense 10 AutoSet for Her. Intervention: Administration of PAP Treatment with suboptimal pressure for 1 night.
  Interventions: Device: AirSense 10 AutoSet for Her

INTERVENTIONS:
Device: AirSense 10 AutoSet for Her — Positive airway pressure

SUMMARY:
The AirSense 10 platform is able to detect respiratory events at night and report these data via telemonitoring. The accuracy of the AirSense 10 will be compared with scoring with polysomnography (PSG). 100 patients will be observed in a sleep facility under PSG and AirSense treatment.

DETAILED DESCRIPTION:
Sleep disordered breathing is commonly assessed by calculating an Apnea-Hypopnea-Index AHI and a Hypopnea-Index HI to define how frequent breathing or breathing efforts stop during the night. The severity of sleep apnea (SA) is determined by the number of occurring apneas and hypopneas. The respiratory disturbance index (RDI) captures these events and is calculated comprising an AHI but also RERAs via the flow signal. Polysomnography (PSG) is being used in the sleep laboratory as the Gold standard method to document a patient's sleep behavior by tracking air flow, respiratory effort, blood oxygen and electrocardiac as well as electromyographic signals. This way a comprehensive sleep pattern analysis can be created and different forms of SA can be detected. However, the method is laborious and cost-intensive, so it could save time and costs to have events accurately scored by the device itself. Device data become important when tracking a patient's sleep night by night and not only once. Reliable sleep data can be a valuable tool for tailoring sleep therapy to specific patient's needs. Accurate device data also build the foundation for analysis of large amounts of data, which can help us understanding how sleep disorders develop.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years who are able to understand and follow the instructions of the study personnel
2. Patients with an indication for PAP therapy or currently adherent to PAP therapy (device usage ≥4 h/ night) for moderate to severe sleep apnoea and diagnostic AHI ˃15/h and/or a residual CAI ˃5/h
3. Patients with currently titrated fixed CPAP pressure ≥8 cmH2O; or 95th percentile APAP pressure ≥8 cmH2O; or ASV therapy with a 95th percentile IPAP of ≥8 cmH2O
4. Patients who are established PAP users (PAP use duration ≥6 weeks)
5. Dated and signed written informed consent

Exclusion Criteria:

1. Patients with moderate to severe obstructive airway disease and/or respiratory insufficiency
2. Patients with heart failure in NYHA class III or IV, unstable hypertension, paroxysmal/persistent atrial fibrillation, unstable angina pectoris, cardiac or cerebral ischemic events within the last 6 months before screening
3. Patients with current primary or secondary insomnia
4. Patients who are pregnant or breastfeeding
5. Patients who are physically unable to comply with the protocol

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the diagnostic accuracy of the AirSense 10 Apnea-Hypopnea-Index (AHI) algorithm compared to polysomnography (PSG) scored AHI. | 1 night
  Calculate accuracy of the device when scoring Apnoeas and Hypopneas by comparing to polysomnography scoring. Identify Apneas (at least 90% decrease of airflow for at least 10 seconds) and Hypopneas (decrease of airflow by at least 30% for at least 10 seconds accompanied by a reduction of Oxygen Saturation of 4%) and calculate the apnea-hypopnea-index (AHI): (apneas + hypopneas)/hours of sleep.

SECONDARY OUTCOMES:
To evaluate the diagnostic accuracy of the AirSense 10 Apnea-Hypopnea-Index (AHI) detection compared to polysomnography (PSG) gold standard scored AHI for clinical relevant threshold values. | 1 night
  For secondary endpoint different cut-off values of AHI will be used to determine the accuracy at clinical relevant thresholds. To calculate device AHI accuracy compared to PSG AHI, receiver-operator-curves will be created and sensitivity and specificity calculated based on an AHI cut-off of 5, 15 or 30.
To evaluate the diagnostic accuracy of the AirSense 10 Obstructive Apnea-Index (OAI) detection compared to polysomnography (PSG) gold standard scored OAI. | 1 night
  Calculate accuracy of the device when scoring obstructive apnoeas by comparing to polysomnography scoring. Identify Apneas (at least 90% decrease of airflow for at least 10 seconds) and calculate the obstructive apnea-index (OAI): (apneas)/hours of sleep.
To evaluate the diagnostic accuracy of the AirSense 10 Central Apnea-Index (CAI) detection compared to polysomnography (PSG) gold standard scored CAI. | 1 night
  Calculate accuracy of the device when scoring central apnoeas by comparing to polysomnography scoring. Identify Apneas (at least 90% decrease of airflow for at least 10 seconds) and calculate the central apnea-index (CAI): (apneas)/hours of sleep.
To evaluate the diagnostic accuracy of the AirSense 10 Respiratory-Disturbance-Index (RDI) detection compared to polysomnography (PSG) gold standard scored RDI. | 1 night
  Calculate accuracy of the device when scoring respiratory disturbances by comparing to polysomnography scoring. Identify Apneas (at least 90% decrease of airflow for at least 10 seconds) and hypopneas (at least 90% decrease of airflow for at least 10 seconds) with a 3%drop in Oxygen saturation from baseline Level, and RERAs (flow Limitation that does not Count as an hypopnea) and calculate the respiratory disturbance-index (RDI): (apneas + hypopneas + RERAs)/hours of sleep.
Evaluate the diagnostic accuracy of the AirSense 10 Respiratory Effort Related Arousals (RERA) detection compared to polysomnography (PSG) gold standard scored RERA. | 1 night
  Calculate accuracy of the device when scoring RERAs by comparing to polysomnography scoring RERAs. Identify RERAs (flow Limitation that does not Count as an hypopnea) and calculate the RERA-Index: RERAs/hours of sleep.
To evaluate the diagnostic accuracy of AirView AHI reporting compared to reporting via ResScan (SD card data) | 1 night
  AirView is a cloud-based ResMed telemonitoring platform where sleep data can be transferred remotely, displayed and analysed. ResScan is an analysis and reporting software, where device data from the memory card is being uploaded.
To evaluate the diagnostic accuracy of AirView RDI reporting compared to reporting via ResScan (SD card data). | 1 night
  AirView is a cloud-based ResMed telemonitoring platform where sleep data can be transferred remotely, displayed and analysed. ResScan is an analysis and reporting software, where device data from the memory card is being uploaded.
Sensitivity, specificity and accuracy of the sleep state detection algorithm of the AirSense10 for Her | 1 night
  Identify the sleep stage: Stage W (wakefulness), stage N1 (NREM1), stage N2 (NREM2), stage N3 (NREM3) and stage R (REM)
Sensitivity, specificity and accuracy of sleep efficiency as derived from the sleep state detection algorithm of the AirSense10 for Her | 1 night
  Calculate sleep efficiency by dividing minutes of sleep by minutes of time in bed

CONTACTS AND LOCATIONS:
Overall Officials: Volker Toepfer, Dr, Principal Investigator — Lungenzentrum Ulm
Locations (2):
- Germany (2):
  - Schlaf- und Beatmungszentrum Blaubeuren, Blaubeuren Abbey, Baden-Wurttemberg
  - Ruhrlandklinik Essen, Essen, North Rhine-Westphalia

REFERENCES:
- [Background] Pepin JL, Guillot M, Tamisier R, Levy P. The upper airway resistance syndrome. Respiration. 2012;83(6):559-66. doi: 10.1159/000335839. Epub 2012 Mar 1. PMID 22377755
- [Background] Berry RB, Budhiraja R, Gottlieb DJ, Gozal D, Iber C, Kapur VK, Marcus CL, Mehra R, Parthasarathy S, Quan SF, Redline S, Strohl KP, Davidson Ward SL, Tangredi MM; American Academy of Sleep Medicine. Rules for scoring respiratory events in sleep: update of the 2007 AASM Manual for the Scoring of Sleep and Associated Events. Deliberations of the Sleep Apnea Definitions Task Force of the American Academy of Sleep Medicine. J Clin Sleep Med. 2012 Oct 15;8(5):597-619. doi: 10.5664/jcsm.2172. PMID 23066376